CLINICAL TRIAL: NCT01917968
Title: A Prospective, Non-Randomized, Parallel Cohort, Multi-center Study of Uphold LITE Versus Native Tissue for the Treatment of Women With Anterior/Apical Pelvic Organ Prolapse
Brief Title: Uphold LITE Post-Market Surveillance Study
Acronym: Uphold LITE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Boston Scientific Corporation (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: U8090
Record Dates: First submitted 2013-07-18; First posted 2013-08-07 (Estimated); Results first posted 2021-03-15 (Actual); Last update posted 2021-05-20 (Actual); Status verified 2021-04

CONDITIONS: Pelvic Organ Prolapse
Keywords: POP; Transvaginal; Native Tissue Repair; Repair Augmented with Mesh; Pelvic Organ Prolapse
MeSH Terms: conditions — Pelvic Organ Prolapse

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Uphold Lightweight Vaginal Support System (Active Comparator): Transvaginal repair with mesh (Uphold LITE)
  Interventions: Device: Uphold Lightweight Vaginal Support System
- Traditional native tissue repair (Active Comparator): Sacrospinous ligament fixation or uterosacral ligament suspension and/or colporrhaphy
  Interventions: Procedure: Traditional native tissue repair

INTERVENTIONS:
Device: Uphold Lightweight Vaginal Support System — Pelvic organ prolapse repair via transvaginal mesh (Uphold LITE)
  Other Names: Uphold LITE
  Arms: Uphold Lightweight Vaginal Support System
Procedure: Traditional native tissue repair — Sarcrospinous ligament fixation or uterosacral ligament suspension and/or colporrhaphy
  Arms: Traditional native tissue repair

SUMMARY:
The purpose of this study is to compare transvaginal mesh repair to traditional native tissue repair in women surgically treated for anterior and/or apical pelvic organ prolapse.

DETAILED DESCRIPTION:
The primary objective is to evaluate clinical effectiveness of transvaginal repair with mesh (Uphold LITE) against traditional native tissue repair in women surgically treated for anterior and/or apical pelvic organ prolapse. Secondary objectives are to evaluate Uphold LITE-related complications and subject reported outcomes.

The primary endpoint of the study is to achieve superiority of transvaginal repair with mesh (Uphold LITE) over native tissue repair at 36 months as compared to baseline. Success will be based on a composite of objective and subjective measures.

Additionally, a co-primary endpoint of the study is to achieve non-inferiority of transvaginal repair with mesh (Uphold LITE) to native tissue repair for safety by comparing rates of serious device or serious procedure related complications between baseline and the 36 month time point.

The secondary endpoints of the study include assessments of complications and subject reported outcomes.

ELIGIBILITY:
Inclusion Criteria:

1. Subject is female
2. Subject is ≥18 years of age
3. Subject has pelvic organ prolapse with the leading edge at or beyond the hymen. At or beyond the hymen is defined as POP-Q scores of Ba≥0 or (for prolapse of the anterior compartment alone) C≥0 (for prolapse of the apical compartment alone) or C≥-1/2 TVL and Ba≥0 (for a multi-compartment prolapse that includes the anterior and apical compartments).
4. Subject reports of a bothersome bulge they can see or feel per PFDI-20, question 3 response of 2 or higher (i.e. responses of "somewhat", "moderately" or "quite a bit")
5. Subject or subject's legally authorized representative must be willing to provide written informed consent
6. Subject is willing and able to comply with the follow-up regimen

Exclusion Criteria:

1. Subject has an active or chronic systemic infection including any gynecologic infection, untreated urinary tract infection (UTI) or tissue necrosis
2. Subject has history of pelvic organ cancer (e.g. uterine, ovarian, bladder, colo-rectal or cervical)
3. Subject has had prior or is currently undergoing radiation, laser therapy, or chemotherapy in the pelvic area
4. Subject has taken systemic steroids (within the last month) or immunosuppressive or immunomodulatory treatment (within the last 3 months)
5. Subject has systemic connective tissue disease (e.g. scleroderma, systemic lupus erythematosus (SLE), Marfans syndrome, Ehlers Danlos, collagenosis, polymyositis polymyalgia rheumatica)
6. Subject has a known neurologic or medical condition affecting bladder function (e.g. multiple sclerosis, spinal cord injury, or stroke with residual neurologic deficit)
7. Subject is seeking obliterative vaginal surgery as treatment for pelvic organ prolapse (colpocleisis)
8. Subject has a previous prolapse repair with mesh in the target compartment
9. Subject is planning to undergo a concomitant repair with use of mesh in the non-target compartment
10. Subject is not able to conform to the modified dorsal lithotomy position
11. Subject has chronic systemic pain that includes the pelvic area or chronic focal pain that includes the pelvis
12. Subject has uncontrolled diabetes mellitus (DM)
13. Subject is currently participating in or plans to participate in another device or drug study during this study
14. Subject has a known hypersensitivity to polypropylene mesh
15. Subject is pregnant or intends to become pregnant during the study

Ages: 18 Years to 100 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 289 (Actual)
Dates: Start 2013-10-10 (Actual); Primary Completion 2020-02-12 (Actual); Study Completion 2020-02-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Karen Noblett, MD, Principal Investigator — University of California, Irvine
Locations (28):
- United States (28):
  - University of Alabama at Birmingham Kirklin Clinic, Birmingham, Alabama
  - Montgomery Women's Health Associates, PC, Montgomery, Alabama
  - UCSD Health/Women's Pelvic Medicine Center, La Jolla, California
  - Sherry Thomas, PC, North Hollywood, California
  - University of CA Irvine Medical Center, Orange, California
  - Kaiser Permanente OB/GYN Urogynecology, San Diego, California
  - Scripps Clinic Carmel Valley, San Diego, California
  - MedStar Washington Hospital Center, Washington D.C., District of Columbia
  - The Florida Bladder Institute, Naples, Florida
  - NorthShore University HealthSystem, Evanston, Illinois
  - Regional Urology, LLC, Shreveport, Louisiana
  - Capital Women's Care - Frederick, Frederick, Maryland
  - Las Vegas Minimally Invasive Surgery Women's Pelvic Health Center, Las Vegas, Nevada
  - Cooper University Hospital, Voorhees Township, New Jersey
  - Columbia University Irving Medical Center/NY Presbyterian Hospital, New York, New York
  - Presbyterian Hospital, Charlotte, North Carolina
  - Lyndhurst Clinical Research, Winston-Salem, North Carolina
  - St. Alexius Medical Center/Mid Dakota Clinic, Bismarck, North Dakota
  - University of Cincinnati Physicians Co, Cincinnati, Ohio
  - Institute for Female Pelvic Medicine & Reconstructive Surgery, Allentown, Pennsylvania
  - Institute for Female Pelvic Medicine & Reconstructive Surgery, North Wales, Pennsylvania
  - Prisma Health System, Greenville, South Carolina
  - Holston Medical Group at Seasons Center for Urogynecology & Advanced Pelvic Surgery, Bristol, Tennessee
  - Dr. M. Mitchell Silver, FACOG, PA, Nacogdoches, Texas
  - Kyle P. McMorries, MD, Nacogdoches, Texas
  - Women's OB/GYN Center, Pasadena, Texas
  - MultiCare Women's Health Care, Covington, Washington
  - Aurora West Allis Medical Center, West Allis, Wisconsin

REFERENCES:
- [Derived] Kahn B, Varner RE, Murphy M, Sand P, Thomas S, Lipetskaia L, Chung DE, Mahdy A, Noblett K. Transvaginal Mesh Compared With Native Tissue Repair for Pelvic Organ Prolapse. Obstet Gynecol. 2022 Jun 1;139(6):975-985. doi: 10.1097/AOG.0000000000004794. Epub 2022 May 2. PMID 35675593

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 337 subjects were screened and 289 subjects were enrolled in the Uphold LITE Postmarket Surveillance Study. 225 subjects were enrolled in the Uphold LITE arm and 64 subjects in the NTR arm. 421 subjects from the AUGS PFD Registry (146 subjects from BSC's Xenform™ 522 study [NCT01945580], 69 subjects from Acell's MatriStem® 522 study, and 206 from Coloplast's 522 Restorelle® study) were pulled into the NTR arm for a total of 485 subjects in the NTR cohort and a total of 710 subjects overall.
Period: Overall Study
Arm/Group | Uphold Lightweight Vaginal Support System | Traditional Native Tissue Repair
Started | 225 | 485
Completed | 171 | 401
Not Completed | 54 | 84
Not completed — Death | 3 | 2
Not completed — Lost to Follow-up | 21 | 39
Not completed — Physician Decision | 1 | 2
Not completed — Withdrawal by Subject | 20 | 35
Not completed — Subject Relocation | 5 | 1
Not completed — 36M Missed Visit | 3 | 2
Not completed — Subject Noncompliance to Scheduled 36M Follow Up Visit | 1 | 0
Not completed — Change in Family Circumstances | 0 | 1
Not completed — No Data Available | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Uphold Lightweight Vaginal Support System | Traditional Native Tissue Repair | Total
Number analyzed (Participants) | 225 | 485 | 710
Age, Continuous [Mean (Standard Deviation); unit: Years] | 66.1 (10.8) | 61.8 (10.5) | 63.2 (10.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 225 | 485 | 710
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 6 | 20 | 26
  Not Hispanic or Latino | 219 | 457 | 676
  Unknown or Not Reported | 0 | 8 | 8
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  White | 210 | 409 | 619
  Asian | 5 | 11 | 16
  Black or African American | 9 | 55 | 64
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 1
  Other | 1 | 6 | 7
  Not disclosed | 0 | 3 | 3
Region of Enrollment [Number; unit: participants]
  United States | 225 | 485 | 710
Smoking [Count of Participants; unit: Participants]
  Current | 18 | 38 | 56
  Previous | 59 | 139 | 198
  Never | 147 | 308 | 455
  Not Recorded | 1 | 0 | 1
Diabetes [Count of Participants; unit: Participants] | 32 | 63 | 95
Menopausal Status [Count of Participants; unit: Participants]
  Premenopausal | 11 | 54 | 65
  Perimenopausal | 5 | 27 | 32
  Postmenopausal | 209 | 404 | 613
Previous Pelvic Surgery [Count of Participants; unit: Participants] | 169 | 235 | 404

OUTCOME MEASURES:

1. Primary Outcome: Primary Efficacy Endpoint - Number of Participants With Composite Anatomic and Symptomatic Success at 36 Months
Description: Success based on a composite of objective and subjective measures:
  1. Objective success was achieved by the subject having an anatomic outcome defined as the leading edge of prolapse at or above the hymen in the operated compartment:
     * Anterior segment: Leading edge of anterior prolapse was at or above the hymen or POP-Q point Ba ≤ 0.
     * Apical segment: The vaginal apex did not descend more than one-half into the vaginal canal (i.e., POP-Q point C < -1/2 TVL) for multi-compartment prolapse or POP-Q point C ≤ 0 for single compartment apical prolapse.
  2. Subjective success was achieved if the patient denied symptoms of vaginal bulging per Pelvic Floor Distress Inventory (PFDI-20) question 3, answering "no" or "yes" but "Not at all" bothersome (< 2).
  3. No retreatment for POP: no additional surgical treatment for POP in the segment(s) of the vagina treated at the index surgery or no pessary use since index surgery (i.e., 'treated segment' refers to the target compartment).
Time Frame: 36 Months
Population: 337 subjects were screened and 289 subjects were enrolled in the Uphold LITE Postmarket Surveillance Study. 225 subjects were enrolled in the Uphold LITE arm and 64 subjects in the NTR arm. 421 subjects from the AUGS PFD Registry (146 subjects from BSC's Xenform™ 522 study [NCT01945580], 69 subjects from Acell's MatriStem® 522 study, and 206 from Coloplast's 522 Restorelle® study) were pulled into the NTR arm for a total of 485 subjects in the NTR cohort and a total of 710 subjects overall.
Measure: Count of Participants; unit: Participants
Arm/Group | Uphold Lightweight Vaginal Support System | Traditional Native Tissue Repair
Number analyzed (Participants) | 225 | 485
Participants
  Intent to Treat Analysis | 201 | 389
  Per Protocol: number analyzed (Participants) | 221 | 480
  Per Protocol | 199 | 384
Statistical Analysis 1: Comparison: Uphold Lightweight Vaginal Support System vs Traditional Native Tissue Repair; Test type: Superiority; p = 0.056, Z statistics — Statistical significance is considered at 0.05 level; P-value is calculated using a Z statistics from the propensity score adjusted estimates. Missing values are handled using multiple imputation; Adjusted difference in percentages = 6.5, 90% CI 2-sided [-0.2 to 13.2]

2. Primary Outcome: Co-Primary Safety Endpoint - Number of Participants With One or More Serious Device-Related and/or Procedure-Related Complications at 36 Months
Description: A co-primary endpoint of the study was to achieve non-inferiority of transvaginal repair with Uphold LITE vs. NTR for safety by comparing the overall complication rate (device-related and/or procedure-related SAEs) at 36 months
Time Frame: 36 months
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Groups:
- Traditional Native Tissue Repair: Sacrospinous ligament fixation or uterosacral ligament suspension and/or colporrhaphy
  Traditional native tissue repair: Sacrospinous ligament fixation or uterosacral ligament suspension and/or colporrhaphy
Arm/Group | Uphold Lightweight Vaginal Support System | Traditional Native Tissue Repair
Number analyzed (Participants) | 225 | 485
Participants
  Intent To Treat Analysis | 7 | 13
  Per Protocol: number analyzed (Participants) | 221 | 480
  Per Protocol | 7 | 12
Statistical Analysis 1: Comparison: Uphold Lightweight Vaginal Support System vs Traditional Native Tissue Repair; Test type: Non-Inferiority — With type I error of 0.05 and type II error of 0.20 (power 80%), 298 subjects (149 subjects per arm) are needed to detect non-inferiority with a margin of 10%; Adjusted difference in percentages = -0.4, 90% CI 2-sided [-2.7 to 1.9] — The propensity score adjusted difference in SAE rate of Uphold LITE transvaginal mesh (TVM) vs. NTR was estimated

3. Secondary Outcome: Secondary Endpoint - Number of Participants With Mesh Erosion and Exposures Over Time in Intent-to-Treat Subjects
Description: Provides a summary of the number of subjects who reported mesh erosion or exposure at each of the study follow-up time points.
Time Frame: 6 Month, 12 Months, 18 Months, 24 Months, 36 Months, Overall
Population: The population includes the 225 subjects in the Transvaginal repair with mesh (Uphold LITE) arm of the study.
Measure: Number; unit: participants
Groups:
- Total: Inclusive
- Mild; Moderate; Severe: Measure of Severity
Arm/Group | Total | Mild | Moderate | Severe
Number analyzed (Participants) | 225 | 225 | 225 | 225
participants
  Erosion : Within 6 Months | 0 | 0 | 0 | 0
  Erosion : Within 12 Months | 0 | 0 | 0 | 0
  Erosion : Within 18 Months | 0 | 0 | 0 | 0
  Erosion : Within 24 Months | 0 | 0 | 0 | 0
  Erosion : Within 36 Months | 0 | 0 | 0 | 0
  Erosion : Overall | 0 | 0 | 0 | 0
  Exposure : Within 6 Months | 3 | 2 | 1 | 0
  Exposure : Within 12 Months | 5 | 4 | 1 | 0
  Exposure : Within 18 Months | 7 | 5 | 2 | 0
  Exposure : Within 24 Months | 8 | 6 | 2 | 0
  Exposure : Within 36 Months | 9 | 7 | 2 | 0
  Exposure : Overall | 11 | 8 | 3 | 0

4. Secondary Outcome: Secondary Endpoint - Number of Participants With One or More Device-Related and/or Procedure-Related Adverse Events
Description: Number of subjects with the following device-related and/or procedure-related adverse events: de novo dyspareunia, pelvic pain, infection, vaginal shortening, atypical vaginal discharge, neuromuscular problems, vaginal scarring, de novo vaginal bleeding, fistula formation, and/or de novo voiding dysfunction. The Intent-to-Treat (ITT) population includes all enrolled subjects who had a surgery initiated; the As Treated population includes all subjects who successfully completed the surgical procedure. Both ITT and As Treated populations are identical to the Overall Number of Participants Analyzed.
Time Frame: 36 Months
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Uphold Lightweight Vaginal Support System | Traditional Native Tissue Repair
Number analyzed (Participants) | 225 | 485
participants
  De novo Dyspareunia : Intent-to-treat | 2 | 6
  De novo Dyspareunia : As treated | 2 | 6
  Pelvic Pain : Intent-to-treat | 11 | 28
  Pelvic Pain : As treated | 11 | 28
  Infection : Intent-to-treat | 23 | 68
  Infection : As treated | 23 | 68
  Vaginal Shortening : Intent-to-treat | 1 | 0
  Vaginal Shortening : As treated | 1 | 0
  Atypical Vaginal Discharge : Intent-to-treat | 2 | 3
  Atypical Vaginal Discharge : As treated | 2 | 3
  Neuromuscular Problems : Intent-to-treat | 10 | 14
  Neuromuscular Problems : As treated | 10 | 14
  Vaginal Scarring : Intent-to-treat | 0 | 1
  Vaginal Scarring : As treated | 0 | 1
  De novo Vaginal Bleeding : Intent-to-treat | 0 | 7
  De novo Vaginal Bleeding : As treated | 0 | 7
  Fistula Formation : Intent-to-treat | 0 | 0
  Fistula Formation : As treated | 0 | 0
  De novo Voiding Dysfunction : Intent-to-treat | 17 | 23
  De novo Voiding Dysfunction : As treated | 17 | 23

5. Secondary Outcome: Secondary Endpoint - PFDI-20 Change From Baseline in Intent-to-Treat Subjects
Description: The Pelvic Floor Distress Inventory-20 (PFDI-20) consists of three components: Pelvic Organ Prolapse Distress Inventory (POPDI; 6 questions), Urinary Distress Inventory (UDI; 6 questions), and Colorectal-Anal Distress Inventory (CRADI; 8 questions). Each individual component score is summed. The total ranges from 0 to 300, with a higher score indicating a greater impact to QOL (i.e., distress symptoms are more noticeable) and a lower score indicating a lesser impact to QOL (i.e., distress symptoms are less noticeable). Reported outcomes are the change from Baseline for the time periods indicated.
Time Frame: 6 Month, 12 Months, 18 Months, 24 Months, 36 Months
Population: 225 Uphold LITE arm subjects and 485 Native Tissue Repair arm subjects had available questionnaire data at Baseline. The number of participants at each follow up time point represents subjects who had available questionnaire data at Baseline and the time point indicated.
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Uphold LITE: Transvaginal repair with mesh (Uphold LITE)
  Uphold Lightweight Vaginal Support System: Pelvic organ prolapse repair via transvaginal mesh (Uphold LITE)
- Native Tissue Repair: Sacrospinous ligament fixation or uterosacral ligament suspension and/or colporrhaphy
  Traditional native tissue repair: Sacrospinous ligament fixation or uterosacral ligament suspension and/or colporrhaphy
Arm/Group | Uphold LITE | Native Tissue Repair
Number analyzed (Participants) | 225 | 485
score on a scale
  6 Months: number analyzed (Participants) | 214 | 443
  6 Months | -78.9 (57.3) | -77.7 (53.2)
  12 Months: number analyzed (Participants) | 203 | 442
  12 Months | -74.8 (61.6) | -76.9 (54.2)
  18 Months: number analyzed (Participants) | 184 | 415
  18 Months | -78.5 (60.9) | -77.3 (53.4)
  24 Months: number analyzed (Participants) | 182 | 417
  24 Months | -81.8 (56.6) | -77.5 (53.9)
  36 Months: number analyzed (Participants) | 170 | 400
  36 Months | -73.5 (59.4) | -77.2 (56.1)

6. Secondary Outcome: Secondary Endpoint - PFIQ-7 Change From Baseline in Intent-to-Treat Subjects
Description: The Pelvic Floor Impact Questionnaire (PFIQ-7) is composed of 3 separate but related assessments: the Urinary Impact Questionnaire, addresses the impact of urinary incontinence symptoms, the Colorectal-Anal Impact Questionnaire addresses the impact of colorectal-anal or bowel symptoms, and the Pelvic Organ Prolapse Impact Questionnaire addresses impact of vaginal and pelvic symptoms. For each question, the low score (0) corresponds to "not at all" and the high score (3) corresponds to "quite a bit". The scores for the UIQ-7, CRAIQ-7 and POPIQ-7 are additive to yield the final PFIQ-7 score, which ranges from 0-300. A lower score means there is a lesser effect on quality of life.
Time Frame: 6 Month, 12 Months, 18 Months, 24 Months, 36 Months
Population: 222 Uphold LITE arm subjects and 485 Native Tissue Repair arm subjects had available questionnaire data at Baseline. The number of participants at each follow up time point represents subjects who had available questionnaire data at Baseline and the time point indicated.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Uphold LITE | Native Tissue Repair
Number analyzed (Participants) | 222 | 485
score on a scale
  6 Months: number analyzed (Participants) | 212 | 443
  6 Months | -51.2 (59.2) | -41.0 (56.1)
  12 Months: number analyzed (Participants) | 200 | 442
  12 Months | -47.7 (66.6) | -41.9 (55.8)
  18 Months: number analyzed (Participants) | 181 | 415
  18 Months | -48.8 (66.4) | -42.9 (58.8)
  24 Months: number analyzed (Participants) | 179 | 417
  24 Months | -50.3 (62.9) | -41.5 (57.6)
  36 Months: number analyzed (Participants) | 167 | 399
  36 Months | -48.1 (62.9) | -41.9 (55.0)

7. Secondary Outcome: Secondary Endpoint - PISQ-12 Change From Baseline in Intent-to-Treat Subjects
Description: The Pelvic Organ Prolapse/Urinary Incontinence Sexual Questionnaire (PISQ-12) is a validated short form that can be used to ascertain improvement in sexual function and desire in women undergoing therapy for pelvic organ prolapse. The PISQ-12 consists of 12 questions graded on a five-point Likert scale ranging from 0 (always) to 4 (never). Values range from 0-48 and a higher score indicates better sexual function. Reported outcomes are the change from Baseline for the time periods indicated.
Time Frame: 6 Month, 12 Months, 18 Months, 24 Months, 36 Months
Population: 90 Uphold LITE arm subjects and 234 Native Tissue Repair arm subjects had available questionnaire data at Baseline. The number of participants at each follow up time point represents those who had available questionnaire data at Baseline and the time point indicated.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Uphold LITE | Native Tissue Repair
Number analyzed (Participants) | 90 | 234
score on a scale
  6 Month: number analyzed (Participants) | 74 | 187
  6 Month | 4.4 (6.2) | 4.4 (6.3)
  12 Month: number analyzed (Participants) | 71 | 191
  12 Month | 3.9 (6.4) | 4.4 (6.3)
  18 Month: number analyzed (Participants) | 62 | 172
  18 Month | 4.1 (5.7) | 4.0 (6.2)
  24 Month: number analyzed (Participants) | 56 | 173
  24 Month | 4.0 (6.2) | 4.6 (6.5)
  36 Month: number analyzed (Participants) | 55 | 156
  36 Month | 4.2 (5.8) | 4.3 (5.8)

8. Secondary Outcome: Secondary Endpoint - TOMUS Pain Score Change From Baseline in Intent-to-Treat Subjects
Description: The TOMUS Pain Score, a visual analog instrument with a scale of 0 (no pain sensation) to 10 (most intense pain sensation imaginable), was used to assess pain associated with surgery for pelvic organ prolapse. There are seven (7) questions each with a maximum score of 10 and a possible score range of 0-70. Reported outcomes are the change from Baseline for the time periods indicated.
Time Frame: 6 Month, 12 Months, 18 Months, 24 Months, 36 Months
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Uphold LITE | Native Tissue Repair
Number analyzed (Participants) | 225 | 485
score on a scale
  6 Months: number analyzed (Participants) | 214 | 443
  6 Months | -3.8 (8.1) | -3.3 (8.3)
  12 Months: number analyzed (Participants) | 203 | 442
  12 Months | -3.4 (8.3) | -3.8 (8.7)
  18 Months: number analyzed (Participants) | 184 | 415
  18 Months | -3.5 (10.6) | -4.2 (9.0)
  24 Months: number analyzed (Participants) | 182 | 417
  24 Months | -3.6 (8.8) | -3.9 (9.1)
  36 Months: number analyzed (Participants) | 170 | 399
  36 Months | -4.3 (8.7) | -4.0 (8.3)

9. Secondary Outcome: Secondary Endpoint: PGI-I for Prolapse Symptoms in Intent-to-Treat Subjects
Description: The Patient Global Impression of Improvement (PGI-I) for prolapse symptoms is a validated QOL instrument that assesses patient perception of overall improvement after surgical interventions for pelvic organ prolapse. The scale is as follows: 1- Very much better; 2- Much better; 3- A little better; 4- No change; 5- A little worse; 6- Much worse; 7- Very much worse.
Time Frame: 6 Month, 12 Months, 18 Months, 24 Months, 36 Months
Population: 289 subjects were enrolled in the Uphold LITE study--225 in the Uphold LITE arm and 64 in the NTR arm. 421 subjects from AUGS PFD Registry (146 subjects from Xenform™ 522 study, 69 subjects from MatriStem® 522 study, and 206 from Restorelle® 522 study) were pulled into the NTR arm for a total of 485 subjects in the NTR cohort and a total of 710 subjects overall. The number of participants for each follow up time point represents subjects who had available questionnaire data at that time point.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Uphold LITE | Native Tissue Repair
Number analyzed (Participants) | 225 | 485
score on a scale
  6 Month: number analyzed (Participants) | 214 | 441
  6 Month | 1.4 (0.7) | 1.3 (0.7)
  12 Month: number analyzed (Participants) | 203 | 442
  12 Month | 1.5 (0.9) | 1.4 (0.9)
  18 Month: number analyzed (Participants) | 184 | 412
  18 Month | 1.4 (0.8) | 1.4 (0.9)
  24 Month: number analyzed (Participants) | 182 | 417
  24 Month | 1.4 (0.9) | 1.4 (0.9)
  36 Month: number analyzed (Participants) | 170 | 399
  36 Month | 1.6 (1.0) | 1.4 (0.9)

10. Secondary Outcome: Secondary Endpoint - Number of Participants With Intervention for Recurrent Prolapse and Complications at 36 Months Post Index Procedure
Description: Compares the office-based and surgical intervention for recurrent prolapse and complications between the Uphold LITE arm and the NTR arm 36 months from the index procedure in the Intent-to-Treat (ITT) and As Treated populations. The ITT population includes all enrolled subjects who had a surgery initiated; the As Treated population includes all subjects who successfully completed the surgical procedure. Both ITT and As Treated populations are identical to the Overall Number of Participants Analyzed.
Time Frame: 36 Months
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Uphold LITE | Native Tissue Repair
Number analyzed (Participants) | 225 | 485
participants
  Office-based Intervention for Recurrence : Intent-to-Treat | 1 | 2
  Office-based Intervention for Recurrence : As Treated | 1 | 2
  Surgical Intervention for Recurrence : Intent-to-Treat | 5 | 15
  Surgical Intervention for Recurrence : As Treated | 5 | 15
  Office-based Intervention for Complications : Intent-to-Treat | 13 | 40
  Office-based Intervention for Complications : As Treated | 13 | 40
  Surgical Intervention for Complications : Intent-to-Treat | 20 | 34
  Surgical Intervention for Complications : As Treated | 20 | 34

11. Secondary Outcome: Secondary Efficacy Endpoint - Number of Participants With Composite Anatomic and Symptomatic Success at 36 Months
Description: Secondary efficacy endpoint defined similarly to the primary efficacy endpoint except for the definition of objective success. Objective success for this endpoint is defined as:
  * Anatomic success in the operated compartment was achieved by:
    * Anterior segment: No anterior prolapse at or beyond the hymen or POP-Q point Ba < 0.
    * Apical segment: The vaginal apex did not descend more than one-half into the vaginal canal (i.e., POP-Q point C < -1/2 TVL) for multi-compartment prolapse or POP-Q point C < 0 for single compartment apical prolapse.
  * Subjective success was achieved if the patient denied symptoms of vaginal bulging per PFDI-20 question 3, answering "no" or "yes" but "Not at all" bothersome (< 2).
  * No retreatment for POP: No additional surgical treatment for POP in segment(s) of the vagina treated at the index surgery or no pessary use since index surgery ('treated segment' refers to the target compartments in this study, which are the anterior and apical compartments).
Time Frame: 36 Months
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Uphold Lightweight Vaginal Support System | Traditional Native Tissue Repair
Number analyzed (Participants) | 225 | 485
Participants
  Intent to treat | 188 | 353
  Per protocol: number analyzed (Participants) | 221 | 480
  Per protocol | 185 | 346

ADVERSE EVENTS:
Time Frame: 36 Months
Arm/Group | Uphold Lightweight Vaginal Support System | Traditional Native Tissue Repair
All-Cause Mortality (participants affected / at risk) | 3/225 | 2/485
Serious Adverse Events (participants affected / at risk) | 12/225 | 27/485
Other Adverse Events (participants affected / at risk) | 108/225 | 312/485
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Uphold Lightweight Vaginal Support System (N=225) | Traditional Native Tissue Repair (N=485)
Cardiac Event- New (Cardiac disorders) | 0 (0) | 6 (6)
Cardiac Event- Worsening (Cardiac disorders) | 0 (0) | 1 (1)
Constipation - Worsening (Gastrointestinal disorders) | 0 (0) | 1 (1)
Ileus / Bowel Obstruction (Gastrointestinal disorders) | 0 (0) | 4 (4)
Other, Specify (Gastrointestinal disorders) | 0 (0) | 1 (1)
Death (General disorders) | 2 (2) | 0 (0)
Fever (General disorders) | 1 (1) | 0 (0)
Infection- Other, Specify Type (General disorders) | 1 (1) | 0 (0)
Infection - Other, specify type (Infections and infestations) | 0 (0) | 4 (6)
Pelvic Infection / Abscess (Infections and infestations) | 0 (0) | 2 (2)
Pulmonary Event, Specify - NEW (Infections and infestations) | 0 (0) | 1 (1)
Urinary Tract Infection (UTI), Lower (Infections and infestations) | 0 (0) | 2 (2)
Ureteral Kink / Injury (Injury, poisoning and procedural complications) | 1 (1) | 2 (2)
Visceral Organ Injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Other, Specify (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Mesh Exposure in Vagina (Product Issues) | 1 (1) | 0 (0)
Hematoma - Retropubic (Renal and urinary disorders) | 0 (0) | 1 (1)
Mixed Incontinence (Renal and urinary disorders) | 1 (1) | 0 (0)
Pelvic Pain - NEW (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Prolapse (Reproductive system and breast disorders) | 2 (2) | 0 (0)
Pulmonary Event, Specify - Worsening (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (2)
Other, Specify (Surgical and medical procedures) | 0 (0) | 1 (1)
Bleeding (Vascular disorders) | 1 (1) | 0 (0)
Bleeding Requiring Blood Transfusion (Vascular disorders) | 1 (1) | 0 (0)
Malignant Hypertension (Vascular disorders) | 1 (1) | 0 (0)
Thrombotic Event (Vascular disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Uphold Lightweight Vaginal Support System (N=225) | Traditional Native Tissue Repair (N=485)
Cardiac Event - NEW (Cardiac disorders) | 0 (0) | 1 (1)
Cardiac Worsening (Cardiac disorders) | 0 (0) | 1 (1)
Constipation - NEW (Gastrointestinal disorders) | 4 (4) | 12 (12)
Constipation - Worsening (Gastrointestinal disorders) | 2 (2) | 5 (5)
Fecal Incontinence - NEW (Gastrointestinal disorders) | 0 (0) | 18 (18)
Fecal Incontinence - Worsening (Gastrointestinal disorders) | 0 (0) | 6 (6)
Hematoma - Retroperitoneal (Gastrointestinal disorders) | 2 (2) | 1 (1)
Hemorrhoids (Gastrointestinal disorders) | 0 (0) | 3 (3)
Ileus / Bowel Obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 2 (2) | 0 (0)
Neuromuscular Disorder, specify type (Gastrointestinal disorders) | 0 (0) | 8 (8)
Other, Specify (Gastrointestinal disorders) | 1 (1) | 7 (7)
Inflammation (General disorders) | 1 (1) | 1 (1)
Neuromuscular Disorder, specify type (General disorders) | 0 (0) | 1 (1)
Other, Specify (General disorders) | 1 (1) | 2 (2)
Pain, Other (General disorders) | 5 (5) | 3 (3)
Infection - Other, specify type (Infections and infestations) | 4 (4) | 9 (10)
Other, Specify (Infections and infestations) | 0 (0) | 1 (1)
Pelvic Infection / Abscess (Infections and infestations) | 2 (2) | 3 (3)
Pulmonary Event, Specify - NEW (Infections and infestations) | 0 (0) | 2 (2)
Upper Respiratory Infection (Infections and infestations) | 0 (0) | 1 (1)
Urinary Tract Infection (UTI), Lower (Infections and infestations) | 31 (43) | 118 (164)
Vaginal Infection (Infections and infestations) | 4 (4) | 16 (18)
Fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (2)
Other, Specify (Injury, poisoning and procedural complications) | 0 (0) | 3 (3)
Visceral Organ Injury (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Buttock Pain (Musculoskeletal and connective tissue disorders) | 4 (4) | 2 (2)
Neuromuscular Disorder, specify type (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1)
Neoplasia, Non-Pelvic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Neuromuscular Disorder, specify type (Nervous system disorders) | 9 (9) | 6 (6)
Neurovascular Event (Nervous system disorders) | 0 (0) | 1 (1)
Mesh Exposure in Vagina (Product Issues) | 10 (12) | 0 (0)
Suture Exposure in Vagina (Product Issues) | 0 (0) | 19 (20)
Difficulty Emptying Bladder - NEW (Renal and urinary disorders) | 13 (13) | 24 (25)
Difficulty Emptying Bladder - Worsening (Renal and urinary disorders) | 1 (1) | 4 (4)
Dysuria (Renal and urinary disorders) | 1 (1) | 4 (7)
Mixed Incontinence- Worsening (Renal and urinary disorders) | 1 (1) | 0 (0)
Mixed Urinary Incontinence (Renal and urinary disorders) | 0 (0) | 1 (1)
Other, Specify (Renal and urinary disorders) | 1 (1) | 5 (5)
Overactive Bladder (Renal and urinary disorders) | 5 (5) | 6 (6)
Stress Incontinence - NEW (Renal and urinary disorders) | 7 (7) | 6 (6)
Stress Incontinence - Worsening (Renal and urinary disorders) | 3 (3) | 21 (21)
Urge Incontinence - NEW (Renal and urinary disorders) | 8 (8) | 8 (8)
Urge Incontinence - Worsening (Renal and urinary disorders) | 1 (1) | 25 (26)
Urinary Frequency (Renal and urinary disorders) | 1 (1) | 6 (6)
Urinary Urgency (Renal and urinary disorders) | 2 (2) | 5 (5)
Weak Urinary Stream (Renal and urinary disorders) | 0 (0) | 1 (1)
Dyspareunia - NEW (De Novo) (Reproductive system and breast disorders) | 3 (3) | 11 (11)
Dyspareunia - Worsening (Reproductive system and breast disorders) | 0 (0) | 3 (3)
Hematoma - Vaginal (Reproductive system and breast disorders) | 1 (1) | 1 (1)
Other, Specify (Reproductive system and breast disorders) | 2 (2) | 4 (4)
Pelvic Pain - New (Reproductive system and breast disorders) | 14 (14) | 39 (41)
Pelvic Pain - Worsening (Reproductive system and breast disorders) | 1 (1) | 2 (2)
Prolapse (Reproductive system and breast disorders) | 20 (20) | 88 (93)
Sensation Of Bulge (Reproductive system and breast disorders) | 26 (27) | 53 (55)
Sensation Of Pressure (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Vaginal Atrophy (Reproductive system and breast disorders) | 0 (0) | 3 (3)
Vaginal Bleeding, De Novo (Reproductive system and breast disorders) | 0 (0) | 9 (10)
Vaginal Discharge, Atypical (Reproductive system and breast disorders) | 2 (2) | 3 (3)
Vaginal Scarring (Reproductive system and breast disorders) | 0 (0) | 2 (2)
Vaginal Shortening (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Vaginal Wall Dehiscence (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Vulvar Itching (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Vulvar Lesion (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Other, Specify (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Lichen Sclerosus (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Skin Condition (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Tissue Granulation (Skin and subcutaneous tissue disorders) | 2 (2) | 33 (33)
Bleeding (Vascular disorders) | 0 (0) | 1 (1)
Hematoma - Other (Vascular disorders) | 0 (0) | 1 (1)
Other, Specify (Vascular disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Before publishing, Institution and Investigator shall submit copies of any proposed publication or presentation to Sponsor for review at least sixty (60) days in advance of submission for publication or presentation to a publisher or other third party. Sponsor reserves the right to delete any Confidential Information or other proprietary information of Sponsor (including trade secrets but not including Results) from the proposed publication or presentation.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-02-28): https://cdn.clinicaltrials.gov/large-docs/68/NCT01917968/Prot_SAP_000.pdf